CLINICAL TRIAL: NCT00852579
Title: Effects of Macrolides on Asthma Control, Airway Inflammation and Bacterial Colonisation in Smokers With Asthma.
Brief Title: Effects of Macrolides on Asthma Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Euan J Cameron (Other)
Collaborators: University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Euan J Cameron, Clinical Research Fellow - Respiratory Medicine, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR010; EUDRACT 2008-007240-34; MRC Grant G0701626; NRES 09/S0703/23
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: Asthma; Smoker; Macrolide
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active treatment.
  Interventions: Drug: Azithromycin
- 2 (Placebo Comparator): Placebo control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Daily dose 250mg
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Asthma is a common disease in Westernised societies, affecting up to 10% of the population. Corticosteroids are the most effective treatment for asthma but the therapeutic response varies considerably between individuals. A major cause of corticosteroid insensitivity in asthma is cigarette smoking. Active cigarette smoking occurs in over 25% of adults with asthma and a further 25% are ex-smokers. In a series of proof of concept clinical studies the investigators demonstrated for the first time that the efficacy of inhaled and oral corticosteroids is markedly impaired in smokers with asthma and to a lesser extent in ex-smokers with asthma. Active cigarette smoking has other detrimental effects on asthma morbidity including more severe symptoms, increased rates of hospitalisation, and accelerated decline in lung function. Smoking cessation advice is often ineffective because many adult smokers with asthma do not believe that they are personally at risk from their smoking, take many years until stopping smoking and frequently restart smoking after quitting. Alternative or additional drugs to corticosteroids are needed for smokers with asthma who are unable to obtain the clinical benefits associated with stopping smoking. In a proof of concept clinical trial the investigators will test the hypothesis that macrolides improve asthma control and reduce sputum neutrophil counts of smokers with chronic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Age 18-70
* Current smoker
* Duration of symptoms >1yr with stability for 4 weeks
* Able to maintain asthma without exacerbations during run in period
* Able to wean off other asthma medication

Exclusion Criteria:

* Ex-smokers or never smokers
* Planning to quit smoking during duration of trial
* Patients with unstable asthma
* Patients with current epilepsy, psychosis or history of significant atrial or ventricular tachyarrhythmia
* Corrected QT-interval greater than 450msec in women, 430msec in men
* Low potassium levels. If can be corrected then screening can continue with confirmation of normal levels prior to taking study medication
* Liver disease (ALT and/or AST levels 2 or more times ULN)
* Significant renal disease (Creatinine or urea levels 2 or more times ULN)
* Any previous severe adverse reactions to macrolides
* Patients who are known to have specific IgE sensitivity or skin test positivity to grass pollen and a history of worsening of asthma due to hay fever will not be recruited from mid May to the end of July
* Upper or lower respiratory tract infection in the 4 weeks prior to randomisation. Run in period can be prolonged in this situation to have 4 weeks with no respiratory infection prior to randomisation.
* Patients who require medications known to interact with azithromycin
* On other immunosuppressants or chronic antibiotics
* Weight less than 45kg
* Frequent asthma exacerbations (greater than 4) requiring oral corticosteroids in the year prior to randomisation
* Current or past diagnosis of allergic-bronchopulmonary-aspergillosis
* Pregnancy and breast feeding
* Mental impairment or language difficulties that makes informed consent not possible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate. | 12 weeks

SECONDARY OUTCOMES:
Spirometry | 12 weeks
Asthma control score | 12 weeks
Average of last 7 days PEF measurements | 12 weeks
Sputum cell counts | 12 weeks
Fraction of expired nitric oxide | 12 weeks
Airway responsiveness to methacholine | 12 weeks
Exacerbation rates | 12 weeks
Cough score | 12 weeks
Diary symptom score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Thomson, FRCP, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Gartnavel General Hospital, Glasgow
  - Crosshouse Hospital, Kilmarnock

REFERENCES:
- [Background] Thomson NC, Chaudhuri R, Livingston E. Asthma and cigarette smoking. Eur Respir J. 2004 Nov;24(5):822-33. doi: 10.1183/09031936.04.00039004. PMID 15516679
- [Background] Richeldi L, Ferrara G, Fabbri LM, Lasserson TJ, Gibson PG. Macrolides for chronic asthma. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD002997. doi: 10.1002/14651858.CD002997.pub3. PMID 16235309
- [Derived] Cameron EJ, Chaudhuri R, Mair F, McSharry C, Greenlaw N, Weir CJ, Jolly L, Donnelly I, Gallacher K, Morrison D, Spears M, Evans TJ, Anderson K, Thomson NC. Randomised controlled trial of azithromycin in smokers with asthma. Eur Respir J. 2013 Nov;42(5):1412-5. doi: 10.1183/09031936.00093913. Epub 2013 Sep 13. No abstract available. PMID 24036246